CLINICAL TRIAL: NCT05425446
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate The Safety, Tolerability, Pharmacokinetics, and Biomarkers of DONQ52 in Celiac Disease Patients (LILY Study)
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics and Biomarker of DONQ52 in Celiac Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DQB101US
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- SAD Cohort 1 (Experimental): All randomized patients will receive one dose of either DONQ52 Dose A or placebo
  Interventions: Drug: DONQ52; Drug: Placebo
- SAD Cohort 2 (Experimental): All randomized patients will receive one dose of either DONQ52 Dose B or placebo
  Interventions: Drug: DONQ52; Drug: Placebo
- SAD Cohort 3 (Experimental): All randomized patients will receive one dose of either DONQ52 Dose C or placebo
  Interventions: Drug: DONQ52; Drug: Placebo
- SAD Cohort 4 (Experimental): All randomized patients will receive one dose of either DONQ52 Dose D or placebo
  Interventions: Drug: DONQ52; Drug: Placebo
- MAD Cohort 1 (Experimental): All randomized patients will receive multiple dose of either DONQ52 Dose E or placebo
  Interventions: Drug: DONQ52; Drug: Placebo
- MAD Cohort 2 (Experimental): All randomized patients will receive multiple dose of either DONQ52 Dose F or placebo
  Interventions: Drug: DONQ52; Drug: Placebo
- MAD Cohort 3 (Experimental): All randomized patients will receive multiple dose of either DONQ52 Dose G or placebo
  Interventions: Drug: DONQ52; Drug: Placebo

INTERVENTIONS:
Drug: DONQ52 — Subcutaneous (SC) injection
Drug: Placebo — Subcutaneous (SC) injection

SUMMARY:
This study is to characterize the safety and tolerability of an investigational drug called DONQ52 and consists of a single ascending dose part (Part A) and a multiple ascending dose part (Part B) in well-controlled celiac disease patients.

ELIGIBILITY:
Inclusion Criteria:

* History of medically diagnosed celiac disease based on biopsies and positive celiac serology.
* Be on a GFD for at least 12 months
* HLA-DQ2.5 genotype
* Experienced at most mild symptoms of celiac disease

Exclusion Criteria:

* Refractory celiac disease
* Positive for any of the 3 serology (-Tissue transglutaminase-2,- Deamidated gliadin peptide-IgA, and deamidated gliadin peptide-IgG)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or higher | Up to 246 days
  Incidence and severity of TEAEs and its relationship to the study drugs
Safety as assessed by Vital signs (blood pressure, body temperature, pulse rate, respiratory rate, percutaneous oxygen saturation) | Up to 246 days
  Abnormality in vital signs
Safety as assessed by Electrocardiograms (ECGs; QT interval, heart rate) | Up to 246 days
  Abnormality in Electrocardiograms (ECGs)
Safety as assessed by Laboratory tests (hematology, blood chemistry, coagulation and urinalysis) | Up to 246 days
  Incidence of laboratory abnormalities, based on clinical laboratory tests

SECONDARY OUTCOMES:
Pharmacokinetics; Serum DONQ52 concentration | Up to 246 days
  Serum DONQ52 concentrations over time
Pharmacokinetics; Maximum serum concentration [Cmax] | Up to 246 days
  Cmax of DONQ52
Pharmacokinetics; Time to maximum serum concentration [Tmax] | Up to 246 days
  Tmax of DONQ52
Pharmacokinetics; Area under the serum concentration time curve [AUC] | Up to 246 days
  AUC of DONQ52
Pharmacokinetics; Half life [T1/2] | Up to 246 days
  T1/2 of DONQ52
Immunogenicity | Up to 246 days
  Prevalence and incidence of anti-drug antibodies (ADAs) to DONQ52

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (21):
- United States (18):
  - Pinnacle Research Group, Anniston, Alabama
  - Mountain View Clinical Research, Denver, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Site Partners, Leesburg, Florida
  - Clinical Site Partners - Orlando, Winter Park, Florida
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Tandem Clinical Research, Marrero, Louisiana
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Columbia University Medical Center, New York, New York
  - Lucas Research - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Aventiv Research, Inc., Columbus, Ohio
  - Digestive Specialists Inc, Dayton, Ohio
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - Alliance for Multispecialty Research, Knoxville, Tennessee
  - Digestive Research of Central Texas, Waco, Texas
  - Care Access Research, Ogden, Utah
- Australia (3):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - University of Sunshine Coast Clinical Trials Centre - Morayfield, Morayfield, Queensland
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).